CLINICAL TRIAL: NCT00226447
Title: A Study on the Viral Kinetics of Different Regimens of Pegylated Interferon and Lamivudine Combination Therapy in HBeAg Positive Chronic Hepatitis B
Brief Title: Different Regimens of Pegylated Interferon and Lamivudine Combination Therapy in Chronic Hepatitis B Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Collaborators: Hoffmann-La Roche (Industry); GlaxoSmithKline (Industry)
Responsible Party: Professor LY Chan, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P03227
Record Dates: First submitted 2005-09-23; First posted 2005-09-27 (Estimated); Last update posted 2008-10-24 (Estimated); Status verified 2008-10

CONDITIONS: Chronic Hepatitis B
Keywords: Chronic Hepatitis B; Pegylated Interferon; Lamivudine
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — Lamivudine

INTERVENTIONS:
Drug: Pegylated Interferon
Drug: Lamivudine

SUMMARY:
The aim is to investigate the best treatment regime of PEG-Intron A and lamivudine combination in terms of viral clearance in chronic hepatitis B patients.

DETAILED DESCRIPTION:
Chronic hepatitis B is a major cause of mortality and morbidity in Hong Kong and most Southeast Asian countries. The efficacy interferon-alfa (IFN-alfa) or lamivudine monotherapy is far from satisfactory with approximately 20% sustained viral response. Extended use of lamivudine is associated with the emergence of drug resistance mutants. As interferon is an immune modulator and lamivudine directly suppresses viral replication, it is therefore logical to combine the 2 drugs for more efficient viral clearance.

Previous studies on IFN-alfa and lamivudine combination treatment of chronic hepatitis B showed marginal benefit over lamivudine monotherapy. In these studies, lamivudine was either started 8 weeks prior to IFN-alfa or simultaneous with IFN-alfa. Recently, we have performed a study comparing the efficacy of polyethylene glycol-interferon alfa-2b (PEG-Intron A) and lamivudine versus lamivudine monotherapy for 1 year in the treatment of chronic hepatitis B. In our protocol, PEG-Intron A is started 8 weeks before the commencement of lamivudine, and PEG-Intron A is given for 32 weeks while lamivudine is given for a total of 52 weeks. Our published results suggested PEG-Intron A and lamivudine combination treatment is far superior to lamivudine monotherapy (end of treatment virological response 92% vs 20%, p=0.0015). We are not certain whether the benefit of PEG-Intron A and lamivudine combination in our study is due to our staggered regime, the superiority of PEG-Intron A over IFN-alfa, or both. The aim of this study is to investigate the best treatment regime of PEG-Intron A and lamivudine combination in terms of viral clearance.

ELIGIBILITY:
Inclusion Criteria:

* HBsAg positive for at least 6 months prior to screening
* Serum HBV-DNA > 10^6 copies per ml at screening
* Serum HBeAg positive at screening
* Abnormal ALT (1.3-10x upper limit normal) within one month prior to entry
* Compensated liver disease with the following minimum criteria:

  1. Hemoglobin within range & not less than 10% from lower normal limit
  2. WBC >= 4,000/mm3
  3. Platelets >= 100,000/mm3
  4. Bilirubin normal (except for Gilbert's disease).
  5. Albumin stable and normal
* Serum creatinine normal or not more than 10% above the upper normal limit
* Thyroid Stimulating Hormone (TSH) within normal limits (Patients requiring medication to maintain TSH levels in the normal range are eligible if all other inclusion/exclusion criteria are met.)
* Alfa-fetoprotein in normal range (obtained within the previous year, or if elevated and < 500 ng/ml with a negative ultrasound for hepatocellular carcinoma at screening).
* Written informed consent

Exclusion Criteria:

* Co-infection with hepatitis C virus and/or HIV
* Evidence or history of decompensated liver disease

  1. Child's B cirrhosis
  2. Ascites, bleeding varices, spontaneous encephalopathy
  3. Hypersplenism (hemoglobin, white cell count, platelet outside inclusion criteria)
  4. Coagulopathy (PT > 13 sec)
* Any known pre-existing medical condition that could interfere with the patient's participation in and completion of the treatment such as:
* Pre-existing psychiatric condition, especially severe depression, or a history of severe psychiatric disorder.
* Patients on anti-depressant therapy are excluded
* CNS trauma or active seizure disorders requiring medication
* Poorly controlled diabetes mellitus
* Immunologically mediated disease (e.g., inflammatory bowel disease (Crohn's disease, ulcerative colitis, idiopathic thrombocytopenic purpura, lupus erythematous, autoimmune hemolytic anemia, scleroderma, severe psoriasis, rheumatoid arthritis).
* Clinical gout
* ANA > 1:320
* documentation that women of childbearing potential are using contraception. A serum pregnancy test obtained within two weeks prior to initiation of treatment must be negative. Female patients must not be breast feeding.
* Any known history of hypersensitivity to nucleoside analogues or interferon
* Previous use of interferon, lamivudine, immunosuppressive drugs or corticosteroid
* Subjects with clinically significant retinal abnormality
* Substance abuse, such as alcohol (>80 g/day), iv drugs and inhaled drugs. If the subject has a history of substance abuse, to be considered for inclusion into the protocol, the subject must have abstained from using the abused substance for at least 2 years. Subjects receiving methadone within the past 2 years are also excluded.
* Subjects not willing to be counseled/abstain from the consumption of alcohol

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30
Dates: Start 2002-12; Primary Completion 2006-07 (Actual); Study Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
HBV DNA reduction at week 52

SECONDARY OUTCOMES:
Normalization of ALT & negative HBV DNA at EOT, negative HBV DNA at EOT & 24 weeks after cessation of treatment, normalization of ALT at the end of treatment and 24 weeks after the cessation of treatment, Safety of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Henry LY Chan, MD, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Cheng Suen Man Shook Hepatitis Center, Institute of Digestive Disease, The Chinese University of Hong Kong, Prince of Wales Hospital, Hong Kong SAR, China

REFERENCES:
- [Background] Lok AS, Wu PC, Lai CL, Lau JY, Leung EK, Wong LS, Ma OC, Lauder IJ, Ng CP, Chung HT. A controlled trial of interferon with or without prednisone priming for chronic hepatitis B. Gastroenterology. 1992 Jun;102(6):2091-7. doi: 10.1016/0016-5085(92)90337-x. PMID 1587429
- [Background] Lai CL, Chien RN, Leung NW, Chang TT, Guan R, Tai DI, Ng KY, Wu PC, Dent JC, Barber J, Stephenson SL, Gray DF. A one-year trial of lamivudine for chronic hepatitis B. Asia Hepatitis Lamivudine Study Group. N Engl J Med. 1998 Jul 9;339(2):61-8. doi: 10.1056/NEJM199807093390201. PMID 9654535
- [Background] Leung NW, Lai CL, Chang TT, Guan R, Lee CM, Ng KY, Lim SG, Wu PC, Dent JC, Edmundson S, Condreay LD, Chien RN; Asia Hepatitis Lamivudine Study Group. Extended lamivudine treatment in patients with chronic hepatitis B enhances hepatitis B e antigen seroconversion rates: results after 3 years of therapy. Hepatology. 2001 Jun;33(6):1527-32. doi: 10.1053/jhep.2001.25084. PMID 11391543
- [Background] Schalm SW, Heathcote J, Cianciara J, Farrell G, Sherman M, Willems B, Dhillon A, Moorat A, Barber J, Gray DF. Lamivudine and alpha interferon combination treatment of patients with chronic hepatitis B infection: a randomised trial. Gut. 2000 Apr;46(4):562-8. doi: 10.1136/gut.46.4.562. PMID 10716688
- [Background] Barbaro G, Zechini F, Pellicelli AM, Francavilla R, Scotto G, Bacca D, Bruno M, Babudieri S, Annese M, Matarazzo F, Di Stefano G, Barbarini G; Lamivudine Italian Study Group Investigators. Long-term efficacy of interferon alpha-2b and lamivudine in combination compared to lamivudine monotherapy in patients with chronic hepatitis B. An Italian multicenter, randomized trial. J Hepatol. 2001 Sep;35(3):406-11. doi: 10.1016/s0168-8278(01)00145-3. PMID 11592603
- [Background] Tsiang M, Rooney JF, Toole JJ, Gibbs CS. Biphasic clearance kinetics of hepatitis B virus from patients during adefovir dipivoxil therapy. Hepatology. 1999 Jun;29(6):1863-9. doi: 10.1002/hep.510290626. PMID 10347131